CLINICAL TRIAL: NCT06903702
Title: A Randomized, Multicenter, Phase II Study of Maintenance Azacitidine and Venetoclax Versus an Allogeneic Stem Cell Transplant in Older Patients (65 Years and Older) With Acute Myeloid Leukemia Who Achieve an MRD Negative Complete Remission After Induction With Azacitidine and Venetoclax
Brief Title: A Study of Azacitidine and Venetoclax Versus a Stem Cell Transplant in People 65 Years and Older With Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-063
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Azacitidine; Venetoclax; Allogeneic Stem Cell Transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Intervention Model Description: This is a randomized, multi-center, open label, phase II study .
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- maintenance arm Azacitidine and Venetoclax (AZA/VEN) (Experimental): Patients randomized to the maintenance arm (AZA/VEN) will be treated with azacitidine given daily for 7 days starting on Day 1 of each Cycle (7 consecutive days or a total of 7 days with a 2 day break due to weekends or holidays is permissible). Venetoclax will be taken orally daily for 28 days. A cycle will be considered 28 days.
  Interventions: Drug: Azacitidine (AZA); Drug: Venetoclax
- Allogeneic hematopoietic stem cell transplantation (Allo-HCT arm) (Experimental): Patients who are randomized to the transplant arm will start the conditioning regimen no later than 6 weeks (day 42) after C2D1 of AZA/VEN.
  Interventions: Procedure: Allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: Azacitidine (AZA) — given daily for 7 days starting on Day 1 of each Cycle
  Arms: maintenance arm Azacitidine and Venetoclax (AZA/VEN)
Drug: Venetoclax — orally daily for 28 days
  Arms: maintenance arm Azacitidine and Venetoclax (AZA/VEN)
Procedure: Allogeneic hematopoietic stem cell transplantation — After the conditioning treatment, the HSCT procedure is part of standard care on Day 0.
  Arms: Allogeneic hematopoietic stem cell transplantation (Allo-HCT arm)

SUMMARY:
The researchers are doing this study to find out if an allogeneic hematopoietic stem cell transplant (HSCT) or maintenance therapy with azacitidine and venetoclax is more effective at keeping AML from coming back (relapsing).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥65 years of age at the time of signing the informed consent form.
* Confirmed diagnosis of acute myeloid leukemia according to the ELN 2017 criteria
* Treatment with azacitidine and venetoclax for the diagnosis of AML

  o The first cycle of study treatment will start 28-42 days after the start of the second cycle of SOC AZA/VEN. In the event that patients can't be admitted for allo-HCT until after Day 42 due to donor related issues, an additional cycle of AZA/VEN will be allowed as a bridge to the transplant, and then initiation of conditioning will start no later than day 42 after the start of the third cycle.
* Patients with adequate organ function to be considered as candidates for allo-HCT:

  * Cardiac: asymptomatic or if symptomatic, then LVEF at rest must be >40% and must improve with exercise.
  * Renal: CrCl ≥50 ml/min (measured or calculated/estimated).
  * Pulmonary: asymptomatic or if symptomatic, DLCO > 50% of predicted (corrected for hemoglobin)
  * Hepatic: < 5x ULN liver function tests and < 2x ULN total serum bilirubin, unless there is congenital benign hyperbilirubinemia.
  * KPS of ≥ 70
* Patients with suitable donor for allo-HCT
* Patients must achieve a morphologic remission <5% blast with MRD negative status by flow cytometry (defined as one or less residual leukemic blasts per 1000 leukocytes (or 10^3)) meeting one of the below:

  * Complete remission (CR) defined as: <5% blasts with ANC> 1000 AND Plt >100K
  * CRh defined as <5% blasts with ANC > 500 AND Plt >50K
  * CRi defined as <5% blasts with ANC< 1000 OR Plt < 100K
* Subject is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Patients who are not considered to be transplant eligible (either due to lack of suitable donor or due to comorbidities/performance status). The reason the patient is not considered transplant eligible will be documented in the eCRF.
* History of prior allo-HCT
* Patients who underwent prior leukemia directed treatment (other than aza/ven)
* Patients with CNS involvement at any time point prior to enrollment.
* Patients with previous exposure to venetoclax or an HMA for the treatment of a myeloid malignancy
* Patients who are planned for treatment other than AZA/VEN
* Patients who are planned for treatment with HMA/VEN with another agent (e.g. a "triplet")
* Presence of any other condition that may increase the risk associated with study participation, and in the opinion of the investigator, would make the patient inappropriate for entry into the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
1-year Relapse free survival (RFS) | 1 year
  Relapse free survival (RFS)- will be defined with patients being alive and without any evidence of disease. i.e. no morphologic relapse and no emergence of minimal residual disease. In the event of emergence of MRD without a morphologic relapse, this will be defined as relapse only if documented on 2 separate time points. For patients alive and in remission at the data cut-off, RFS will be censored at the last assessment date.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  will be defined with patients being alive and non-relapse mortality (NRM) will be defined as death in the absence of disease recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Tamari, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Follow-up), Middletown, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center - Suffolk (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm